CLINICAL TRIAL: NCT06074601
Title: Observational Study of Pregnant People to Validate Biomarkers of Pregnancy Complication Risk
Brief Title: MIRACLE of LIFE Study
Acronym: MoL
Status: Active, not recruiting | Type: Observational
Sponsor: Mirvie (Industry)
Responsible Party: Sponsor
Other Study IDs: MV-001; Pro00050765 (Other: Advarra IRB)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Preterm Labor; Preterm Birth; Preterm Birth Complication; Preterm Premature Rupture of Membrane; Preeclampsia; HELLP; Gestational Hypertension; Gestational Diabetes Mellitus in Pregnancy; Small for Gestational Age at Delivery; Intrauterine Growth Restriction
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth; Preterm Premature Rupture of the Membranes; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant People: Enrolling any pregnant person over the age of 18 with a singleton pregnancy with their pregnancy having been effectively dated by first trimester ultrasound or last menstrual period
  Interventions: Diagnostic Test: Mirvie Predictive Test for Adverse Pregnancy Outcomes

INTERVENTIONS:
Diagnostic Test: Mirvie Predictive Test for Adverse Pregnancy Outcomes — This is a proprietary biomarker and clinical factor-based algorithm for predicting which pregnancies are at greatest risk of developing a variety of adverse pregnancy outcomes (e.g., preterm birth, preeclampsia)

SUMMARY:
The goal of this observational study is to develop and validate cell-free RNA-based biomarkers for predicting a variety of adverse pregnancy outcomes in a pregnant person population. The main question it aims to answer are:

1. Can cell-free RNA-based biomarkers predict which pregnant people are at greatest risk of developing adverse pregnancy outcomes (e.g., preterm birth, preeclampsia)?
2. What is the performance of such biomarkers when predicting an adverse pregnancy outcome (e.g., sensitivity, specificity, PPV, NPV, TPR)?

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational cohort study, that involves the collection of blood samples from pregnant people during their second trimester of pregnancy. Maternal plasma is isolated from blood samples and subjected to transcriptome and other multi-omic analyses. In conjunction with blood sample collection, extensive clinical data are collected about the pregnancy including any pregnancy complications (e.g., preterm birth, preeclampsia) that may have arisen during pregnancy. Biological markers and clinical data are combined to develop and validate Mirvie's investigational predictive test.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide written informed consent.
2. Subject is willing and able to provide up to 40 mL of blood via venipuncture and comply with all other study procedures.
3. Subject is a pregnant female before 22 weeks of gestation
4. Subject is at least 18 years of age

Exclusion Criteria:

1. Estimated due date (EDD) via 1st or 2nd ultrasound, date of last menstrual period (LMP), or in-vitro fertilization (IVF) implantation date is not available
2. Subject is pregnant with multifetal gestation (e.g., twins)
3. Subject is planning to deliver via home birth

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to biological females who are pregnant and identify as female, male, or non-binary
Study Population: This study will enroll a diverse and representative population of pregnant people from across the United States who meet study inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical validation of cell-free RNA-based biomarkers of adverse pregnancy outcomes | December 2024
  This study will measure the test performance (e.g., ROC, sensitivity, specificity, negative and positive predictive value) of cell-free RNA-based biomarkers that are predictive of a variety of adverse pregnancy outcomes (e.g., preterm birth, preeclampsia)

SECONDARY OUTCOMES:
Discovery of multi-omic biomarkers of adverse pregnancy outcomes | December 2026
  This study will enable the identification of other biomarkers (e.g., proteomic, metabolomic) of adverse pregnancy outcomes

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California San Diego, San Diego, California
  - Women's Care Florida, Orlando, Florida
  - Ochsner Health System, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - MultiCare, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers

REFERENCES:
- [Background] Rasmussen M, Reddy M, Nolan R, Camunas-Soler J, Khodursky A, Scheller NM, Cantonwine DE, Engelbrechtsen L, Mi JD, Dutta A, Brundage T, Siddiqui F, Thao M, Gee EPS, La J, Baruch-Gravett C, Santillan MK, Deb S, Ame SM, Ali SM, Adkins M, DePristo MA, Lee M, Namsaraev E, Gybel-Brask DJ, Skibsted L, Litch JA, Santillan DA, Sazawal S, Tribe RM, Roberts JM, Jain M, Hogdall E, Holzman C, Quake SR, Elovitz MA, McElrath TF. RNA profiles reveal signatures of future health and disease in pregnancy. Nature. 2022 Jan;601(7893):422-427. doi: 10.1038/s41586-021-04249-w. Epub 2022 Jan 5. PMID 34987224
- [Background] Camunas-Soler J, Gee EPS, Reddy M, Mi JD, Thao M, Brundage T, Siddiqui F, Hezelgrave NL, Shennan AH, Namsaraev E, Haverty C, Jain M, Elovitz MA, Rasmussen M, Tribe RM. Predictive RNA profiles for early and very early spontaneous preterm birth. Am J Obstet Gynecol. 2022 Jul;227(1):72.e1-72.e16. doi: 10.1016/j.ajog.2022.04.002. Epub 2022 Apr 6. PMID 35398029